CLINICAL TRIAL: NCT03727321
Title: Fecal Microbial Transplantation and Fiber Supplementation in Subjects With Obesity and Metabolic Syndrome
Brief Title: FMT and Fiber in Patients With Metabolic Syndrome
Acronym: FMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: The Weston A. Price Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00076642
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Fecal microbial transplant; obesity; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Dietary Fiber; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo: Placebo will consist of cellulose powder (Microcrystalline cellulose:Blanver) in foil packets.
  Interventions: Dietary Supplement: Cellulose
- Fecal Microbial Transplant and cellulose (Experimental): 1. Fecal Microbial Transplant - Fecal microbiome transplant (FMT): 50grams of FMT from a single, universal donor will be administered in 20-30 capsules taken by mouth.
  2. Cellulose x 6weeks
  Interventions: Combination Product: Fecal Microbial Transplant; Dietary Supplement: Cellulose
- Fiber (Experimental): Soluble corn fiber (PROMITOR®: Tate&Lyle), Resistant Wheat Starch 4 (Fibersym®: MGP Ingredients), Acacia Gum (Pre-Hydrated Gum Arabic: TIC GUMS).
  Interventions: Dietary Supplement: Fiber
- Fecal Microbial Transplant and Fiber (Experimental): 1. Fecal Microbial Transplant
  2. Soluble corn fiber (PROMITOR®: Tate&Lyle), Resistant Wheat Starch 4 (Fibersym®: MGP Ingredients), Acacia Gum (Pre-Hydrated Gum Arabic: TIC GUMS).
  Interventions: Combination Product: Fecal Microbial Transplant; Dietary Supplement: Fiber

INTERVENTIONS:
Combination Product: Fecal Microbial Transplant — Fecal microbiome transplant (FMT): 50grams of FMT from a single, universal donor will be administered in 20-30 capsules taken by mouth.
  Other Names: FMT
  Arms: Fecal Microbial Transplant and Fiber; Fecal Microbial Transplant and cellulose
Dietary Supplement: Fiber — A combination of soluble corn fiber (PROMITOR®: Tate&Lyle), Resistant Wheat Starch 4 (Fibersym®: MGP Ingredients), and Acacia Gum (Pre-Hydrated Gum Arabic: TIC GUMS) for a total of 6 weeks (men 33g/day; women 27g/day)
  Arms: Fecal Microbial Transplant and Fiber; Fiber
Dietary Supplement: Cellulose — Placebo will consist of cellulose powder (Microcrystalline cellulose:Blanver) in foil packets.
  Arms: Fecal Microbial Transplant and cellulose; Placebo

SUMMARY:
This study is looking at the safety and effectiveness of stool transplant, also known as Fecal Microbiota Transplantation (FMT) and prebiotic supplementation in the management of metabolic syndrome.

Metabolic syndrome is a common progressive medical condition that is linked to obesity, diabetes, and heart disease. Obesity and metabolic syndrome are associated with abnormalities in gut flora which lead to chronic inflammation. This chronic inflammation is thought to worsen the insulin resistance and heart disease seen with metabolic syndrome. Current treatment strategies have shown limited effect, are expensive, and have side effects with long-term use.

FMT is a one-time treatment that has been shown to replace the abnormal gut flora and improve metabolic disease by increasing anti-inflammatory short chain fatty acid (SCFA) production. However, the effects from FMT are not permanent. Prebiotic supplementation is one strategy that may help to extend the benefits of FMT by helping sustain high SCFA levels. At this point, it is not known how FMT and prebiotics work together to affect SCFA levels in participants with metabolic syndrome.

This study will look at this interaction and answer if prebiotic therapy is effective in prolonging the benefits of FMT in participants with metabolic syndrome.

DETAILED DESCRIPTION:
3.0 Design This is an exploratory four-arm, parallel design, randomized placebo-controlled intervention study in obese individuals with metabolic syndrome to evaluate whether FMT from lean donors combined with supplementation with prebiotic fiber will have a clinically significant effect on metabolic parameters. The study includes a 2-week screening/baseline period followed by a single FMT and a 6 week study period in which prebiotic fiber or placebo will be added in powdered form to the subject's normal diet for the duration of the trial (Appendix 1). A follow-up visit at 12 weeks will be done to determine if beneficial effects are maintained in the absence of ongoing fiber intake. A parallel arm design was chosen to avoid cross-over effects.

The four groups are:

1. Control (Placebo FMT and cellulose)
2. FMT only (FMT followed by cellulose)
3. Prebiotic only (Placebo FMT and prebiotic fiber)
4. FMT + prebiotic fiber Schedule and Procedures: Subjects will attend a total of 5 clinic appointments throughout the study for anthropometric and blood pressure measurements, dietary intake, hunger and satiety, and quality of life assessment using questionnaires, and for collection of blood and fecal samples (Appendix 2). The intervention will be stopped at 6 weeks. A final follow-up visit will occur at 12 weeks for anthropometric and blood pressure measurements, and collection of blood and stool samples.

3.1 Randomization Subjects will be randomized to one of 4 groups via computer-generated numbers and stratified by gender. Individuals will be blinded as to their group allocation to reduce bias. Randomization concealment will be protected by several levels of security, including our secure website, password protection by only those authorized to randomize and a variable blocked randomization.

3.2 Maintenance

Randomized codes will be maintained in REDCAP. Codes will be broken at the end of the trial.

3.3 Trial Treatment

Fecal microbiome transplant (FMT): 50grams of FMT from a single, universal donor will be administered in 20-30 capsules taken by mouth. These capsules will be frozen at -700C until date of administration on day 1 of the trial. The FMT will be given after individuals have fasted overnight and completes a bowel preparation using Pico-Salax®, a routine colonoscopy preparation. The study will use only one donor to reduce variability in donor profiles unless this donor becomes unavailable at which point backup donors will be available. Placebo FMT will consist of cellulose pills.

Fiber Supplementation:

Soluble corn fiber (PROMITOR®: Tate&Lyle)

* Women: 4.5 gm of PROMITOR by mouth days 1-3 increased to 9 gm daily from day 4 until trial completion.
* Men: 5.5 gm of PROMITOR by mouth days 1-3 increased to 11 gm by mouth daily from day 4 until trial completion.

Resistant Wheat Starch 4 (Fibersym®: MGP Ingredients):

* Women: 4.5 gm of powdered RS4 by mouth days 1-3 increased to 9 gm by mouth daily from day 4 until trial completion.
* Men: 5.5gm of powdered RS4 by mouth days 1-3 increased to 11 gm by mouth daily from day 4 until trial completion.

Acacia Gum (Pre-Hydrated Gum Arabic: TIC GUMS):

* Women: 4.5 gm of powdered acacia gum by mouth days 1-3 increased to 9 gm by mouth daily from day 4 until trial completion.
* Men: 5.5gm of powdered acacia gum by mouth days 1-3 increased to 11 gm by mouth daily from day 4 until trial completion.

The product will be supplied to patients on a weekly basis in pre-weighed foil packets.

Placebo: Placebo will consist of cellulose powder (Microcrystalline cellulose:Blanver) in identical foil packets.

3.4 Duration

The study duration is 12 weeks. Subjects will be seen in the clinic at recruitment, and then at 2 and 6 weeks following FMT. Intervention will be from 1-6 weeks. A final follow-up visit will occur at 12 weeks (Appendix 1)

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 and < 65 years at the time of screening

  * BMI > 30
  * Total body weight fluctuation over the last 6 months less than 10%
  * Fasting plasma glucose > 5.6 mmol/L OR HgbA1c ≥5.5% OR patients receiving an antidiabetic medication
  * At least one of the following:

    * Fasting triglyceride ≥1.7 mmol/L OR receiving dyslipidemia medication
    * HDL cholesterol <1.03 mmol/L in males or <1.29 mmol/L in females OR receiving dyslipidemia medication
    * Known diagnosis of hypertension OR systolic blood pressure ≥130 or diastolic blood pressure ≥85 mmHg OR receiving antihypertension medication

Exclusion Criteria:

* • Systolic blood pressure ≥180 or diastolic blood pressure ≥110 mmHg at screening.

  * Triglyceride ≥6 mmol/L.
  * Acute infectious or inflammatory condition over the presiding 4 weeks.
  * Current or recent use (Previous 6 months) of insulin for diabetes control.
  * History of oropharyngeal or significant esophageal dysphagia, inflammatory bowel disease, colon cancer, or colonic polyps with high grade dysplasia.
  * History of autoimmune conditions or chronic inflammatory condition, such as rheumatoid arthritis, chronic active hepatitis B or C, HIV, chronic pancreatitis, advanced NASH, or liver cirrhosis.
  * Active malignancy.
  * Active substance abuse or excessive EtOH (defined as >2 X 8oz drinks/d).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity Assessment | 12 weeks
  The homeostasis Model Assessment-Insulin Resistance (HOMA-IR) is a mathematical model to predict the interaction between glucose and insulin dynamics across a range of glucose plasma levels assuming a feedback circuit between the liver and β-cells in the pancreas

SECONDARY OUTCOMES:
Health-related quality of life (HRQL): EQ-5D Index | 12 week
  Assessment of the current health related quality of life will be accomplished by conducting standardized interviews and by using the validated questionnaires EQ-5D Index. Participants will report perceived health outcomes using this validated survey, and rank overall perceived health from 0 (low)- 100 (high).
Dietary Intake | 12 week
  Dietary intake will be assessed for each clinic using MyFitnessPal.
Inflammatory markers | 12 week
  . Levels of leptin, ghrelin, adiponectin, TNFα, IL-6, LPS (lipopolysaccharide), LPS-binding protein and zonulin will be determined using currently accepted laboratory techniques.
Stool Microbiome | 12 weeks
  Stool microbiome will be analyzed for Operational Taxonomic Unit determination.
Anthropometric Measurements | 12 weeks
  BMI (kg/m2)
Fasting lipid profile | 12 weeks
  Changes in Fasting lipid profile between baseline and 6 and 12 weeks
Glucose Tolerance Assessment | 12 weeks
  The oral glucose tolerance test (OGTT) is a dynamic test that reflects the efficiency of the body to dispose of glucose after an oral load. It is commonly used in clinical scenarios to diagnose glucose intolerance and diabetes. [33] After overnight fast (> 8 h), blood samples for determination of glucose and insulin concentration will be taken at -5, 0, 30, 60, and 120 min following a standard oral glucose load.
Hunger and Satiety Assessment | 12 weeks
  Assessed via the standardized hunger and satiety questionnaire (categorical variables with no analog scale)
Gastrointestinal tolerance | 12 weeks
  Assessed via the standardized gastrointestinal tolerance questionnaire (categorical variables with no analog scale)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Madsen, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be kept private and not distributed to other researchers outside of our study group. After the study is done, we will keep data stored for 25 years.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03727321/Prot_SAP_000.pdf